CLINICAL TRIAL: NCT06578455
Title: A Randomized, Open-Label, 4-Way Crossover, Pharmacokinetic Study to Compare CBD-NE to Epidyolex in Healthy Adult Volunteers Under Both Fed and Fasted Conditions
Brief Title: A Pharmacokinetic Study to Compare CBD-NE to Epidyolex in Healthy Adult Volunteers Under Both Fed and Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: T0051
Record Dates: First submitted 2024-08-20; First posted 2024-08-29 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-09

CONDITIONS: CBD Pharmacokinetics; Healthy Participants
Keywords: Cannabidiol; Pharmacokinetic; Safety
MeSH Terms: interventions — Cannabidiol; Powders

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, Crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CBD-NE Under Fed Condition (Experimental): A single dose of CBD-NE (6 capsules) following consumption of a high-fat, high-calorie breakfast
  Interventions: Drug: Cannabidiol (CBD) Powder
- TP Under Fasted Condition (Experimental): A single dose of CBD-NE (6 capsules) after a minimum 10-hour fast
  Interventions: Drug: Cannabidiol (CBD) Powder
- Epidyolex Under Fed Condition (Active Comparator): A single dose of Epidyolex (4 mL oil) following consumption of a high-fat, high-calorie breakfast
  Interventions: Drug: Cannabidiol 100 MG/ML [Epidiolex]
- Epidyolex Under Fasted Condition (Active Comparator): A single dose of Epidyolex (4 mL oil) after a minimum 10-hour fast
  Interventions: Drug: Cannabidiol 100 MG/ML [Epidiolex]

INTERVENTIONS:
Drug: Cannabidiol (CBD) Powder — 66.68 mg CBD per capsule for a total of 400 mg CBD per serving
  Other Names: CBD-NE
  Arms: CBD-NE Under Fed Condition; TP Under Fasted Condition
Drug: Cannabidiol 100 MG/ML [Epidiolex] — 100 mg CBD/mL for a total of 400 mg CBD per serving
  Other Names: Epidyolex
  Arms: Epidyolex Under Fasted Condition; Epidyolex Under Fed Condition

SUMMARY:
Cannabidiol (CBD), derived from the Cannabis sativa plant, is being investigated for its potential health benefit without the psychoactive properties and adverse reactions that arise from the use of delta-9-tetrahydrocannabinol (Δ9-THC). Few studies have characterized the pharmacokinetic (PK) effects and safety of oral CBD administration. Epidiolex (Epidyolex), an oil form of CBD, is the only marketed monotherapy approved by the United States Food and Drug Administration (FDA) and Health Canada. Delivery of a CBD in a powder/capsule form may provide a more efficient method for consumers.

The goal of this study is to characterize the PK profile of the test product, CBD-NE (a capsule formulation) compared to Epidyolex under both fasted and fed conditions. Each participant will receive a dose of each product under both fed and fasted conditions in a crossover design.

DETAILED DESCRIPTION:
CBD and Δ9-THC are the most abundant extracts from the Cannabis sativa plant. Δ9-THC is typically associated with psychotropic effects due to its affinity for cannabinoid receptor types 1 and 2. CBD possesses a low affinity and lack of function at these receptors; therefore there is an interest in its potential health benefit without the psychoactive properties and adverse reactions that arise from Δ9-THC use. Only few studies have characterized the PK effects and the safety of oral CBD administration. As CBD is a lipophilic molecule, consuming CBD with a lipid formulation may increase its exposure. Additionally, CBD is known to have poor bioavailability when taken orally because it is rapidly metabolized by the liver to 7-hydroxycannabidiol (7-OH-CBD) and then to cannbidiol-7-oic acid (7-COOH-CBD), which may reduce the potency of CBD. Formulation strategies for orally consumed CBD products are being investigated to by-pass one or both of these limitations and improve the bioavailability of CBD. Epidyolex, a purified form of CBD, is delivered in a solution of sesame oil which aids absorption. Epidyolex, marketed and sold in the US and Canada as Epidiolex, is currently the only marketed CBD monotherapy with US FDA and Health Canada approval and is approved for treatment of certain types of epilepsy. However, administration of CBD in oil form is not ideal for consumers as it is not always convenient or precise. Delivery of CBD in a powder/capsule form may provide a more efficient method of CBD consumption.

The test product will be CBD-NE, a novel formulation of CBD in a powder form. This product will be investigated in healthy adults as its PK profile is not yet characterized in humans. This study is designed to be a randomized, crossover, comparator control trial to evaluate the PK profile and safety of CBD-NE compared to Epidyolex in healthy adults under both fed and fasted conditions.

Two study products, CBD-NE and Epidyolex, will be administered under both fed and fasted conditions. Participants will be randomized in a 1:1:1:1 ratio to one of 4 treatment sequences. There will be a total of 4 treatment periods consisting of 2 consecutive days, and one washout period. Each dose will be followed by a minimum 14-day, maximum of 28-day washout period, with the last dose followed by a follow-up phone call which will occur within the timeframe of the longest washout period over the study. For the fed state, participants will consume a high-fat, high-calorie breakfast within the 30 minutes prior to dosing.

Pharmacokinetic blood sampling will occur pre-dose and at 0.25 h, 0.5 h, 0.75 h, 1.0 h, 1.5 h, 2.0 h, 3.0 h, 4.0 h, 5.0 h, 6.0 h, 8.0 h, 12.0 h and 24.0 h post-dose.

Blood samples collected will be used to assess the PK profiles of CBD-NE and Epidyolex. PK parameters measured will include maximum concentration in plasma (Cmax), time to reach maximum concentration (Tmax), elimination half-life (T1/2), area under the plasma concentration-time curve over 24 hours (AUC0-24), area under the plasma concentration-time curve from zero to infinity (AUCinf) and AUC0-24/AUCinf for CBD, 7-OH-CBD and 7-COOH-CBD. Safety endpoints will be assessed throughout the study and will include reports of adverse events, 12-lead ECG, vital signs, safety laboratory assessments, and abbreviated physical exam.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants who are 19 to 55 years of age (inclusive).
2. Have a body mass index (BMI) range of 18.0 - 29.9 kg/m2 (inclusive) and body weight ≥ 50 kg.
3. In good general health as deemed by the investigator.
4. Naïve to oral or inhaled cannabis or hemp, or light user of oral or inhaled cannabis or hemp products (not more than 2 times per month on average) who have used cannabis for recreational (non-therapeutic) purposes without severe side effects.
5. Non-smoker (including nicotine vaping) and have not used any nicotine products (e.g., patches, gums, etc.) for >3 months prior to the first PK blood draw (Visit 2). Note: A non-smoker is defined as someone who does not habitually/regularly use products containing nicotine.
6. Have suitable veins for repeated venipuncture.
7. Have systolic blood pressure within 90 to 139 mmHg (inclusive) and diastolic blood pressure within 60 to 89 mmHg (inclusive) at screening and Visit 2.
8. Able to consume oil formulation, and swallow pills or capsules whole, and without chewing.
9. Agree to follow the restrictions on concomitant treatments listed in the protocol.
10. Agree to follow the restrictions on lifestyle listed in the protocol.
11. Agree to adhere to the contraception requirements for this study.
12. Able to consume the entire high-fat, high-calorie breakfast provided within 30 minutes at the site during Visits 2 and 4.
13. Agree to fast overnight, i.e., no food or liquids (except for water, permitted up to 1 h prior to dosing) for a minimum 10 h prior to starting the high-fat, high-calorie breakfast on Visits 2 and 4 or prior to dosing on Visits 6 and 8.
14. Have maintained consistent dietary habits (including supplement intake) and lifestyle for the last 3 months prior to screening.
15. Willing and able to agree to the requirements and restrictions of this study, be willing to voluntarily consent, and carry out all study related procedures.

Exclusion Criteria:

1. Participants who are lactating, pregnant, or planning to become pregnant during the study as confirmed by a positive pregnancy test during study visits or not willing to perform a pregnancy test.
2. Male participants that are planning to conceive during the study.
3. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients, or any of the items that could be included in the standardized meals/snacks.
4. Current COVID-19 infection at the time of screening or Visit 2, or currently have the post COVID-19 condition as defined by the World Health Organization (WHO) (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by alternative diagnosis).
5. Presence of any clinically significant or abnormal results from laboratory tests at screening (Visit 1) and/or vital sign assessments at Visits 1 or 2 as judged by the investigator and or/designee.
6. Demonstrates a positive screen for Hepatitis B Surface Antigen (HBsAg), Hepatitis C (HCV), or Human Immune Deficiency Virus (HIV) at screening.
7. Demonstrates a positive urine drug screen, positive cotinine test or positive breath alcohol test at screening or Visit 2.
8. Have abnormal 12-lead electrocardiogram (ECG) results at screening or Visit 2 as determined at the discretion of the investigator.
9. Evidence of hepatic or renal dysfunction as evidenced by alanine aminotransferase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP) or gamma-glutamyl transferase (GGT) being ≥ 2 times the upper limit of normal or serum creatinine value ≥ 176.84 µmol/L at screening.
10. Have thyroid disease, Type I or Type II diabetes.
11. Have a history of blood clotting disorders.
12. Have a history of heart disease/cardiovascular disease, renal or hepatic impairment/ disease, bipolar disorder, immune disorders and/or immunocompromised [(e.g., HIV/acquired immunodeficiency syndrome (AIDS)].
13. Have a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to the screening visit.
14. Have an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea).
15. Have medical condition(s) known to interfere with absorption, distribution, metabolism or excretion of the study product (e.g., Crohn's disease, short bowel, acute or chronic pancreatitis or pancreatic insufficiency).
16. Major surgery with general anesthesia in the 3 months prior to screening or planned major surgery during the study.
17. Reports a significant blood loss or blood donation totaling between 101 mL to 449 mL of blood within 30 days prior to the first PK visit (Visit 2) or a blood donation of more than 450 mL within 56 days prior to Visit 2.
18. Reports donating plasma (e.g., plasmapheresis) within 15 days prior to Visit 2.
19. History of alcohol or substance abuse in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program).
20. Currently consumes, on average, more than 2 standard alcoholic beverages a day or has any habit of alcohol use that, to the opinion of the investigator, may be of a concern for the study. A standard alcoholic beverage is defined as 12 ounces of beer, 5 ounces of wine, or 1.5 ounces of liquor.
21. Receipt or use of test product(s) in another research study within 28 days prior to Visit 2 or longer if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.
22. Any other medical condition/situation or use of medications/supplements/therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Properties of CBD-NE compared to Epidyolex under Fed Conditions | 0-24 hours
  Area under the plasma concentration-time curve over 24 hours (AUC0-24) for CBD
PK Properties of CBD-NE compared to Epidyolex under Fasted Conditions | 0-24 hours
  AUC0-24 for CBD

SECONDARY OUTCOMES:
PK Properties of CBD-NE compared to Epidiolex under Fed Conditions | 0-24 hours
  AUC0-24 for 7-hydroxycannabidiol (7-OH-CBD) and cannabidiol-7-oic acid (7-COOH-CBD)
PK Properties of CBD-NE compared to Epidyolex under Fasted Conditions | 0-24 hours
  AUC0-24 for 7-OH-CBD and 7-COOH-CBD
PK Properties of CBD-NE compared to Epidyolex under Fed Conditions | 0-24 hours
  Maximum concentration in plasma (Cmax) for CBD, 7-OH-CBD and 7-COOH-CBD
PK Properties of CBD-NE compared to Epidyolex under Fasted Conditions | 0-24 hours
  Cmax for CBD, 7-OH-CBD and 7-COOH-CBD
PK Properties of CBD-NE compared to Epidyolex under Fed Conditions | 0-24 hours
  Time to reach Cmax (Tmax) for CBD, 7-OH-CBD and 7-COOH-CBD
PK Properties of CBD-NE compared to Epidyolex under Fasted Conditions | 0-24 hours
  Tmax for CBD, 7-OH-CBD and 7-COOH-CBD
PK Properties of CBD-NE compared to Epidyolex under Fed Conditions | 0-24 hours
  Elimination half-life (T1/2) for CBD, 7-OH-CBD and 7-COOH-CBD
PK Properties of CBD-NE compared to Epidyolex under Fasted Conditions | 0-24 hours
  T1/2 for CBD, 7-OH-CBD and 7-COOH-CBD
PK Properties of CBD-NE compared to Epidyolex under Fed Conditions | 0-24 hours
  Area under the plasma concentration-time curve from zero to infinity (AUCinf) for CBD, 7-OH-CBD and 7-COOH-CBD
PK Properties of CBD-NE compared to Epidyolex under Fasted Conditions | 0-24 hours
  AUCinf for CBD, 7-OH-CBD and 7-COOH-CBD
PK Properties of CBD-NE compared to Epidyolex under Fed Conditions | 0-24 hours
  Ratio of AUC0-24 to AUCinf for CBD, 7-OH-CBD and 7-COOH-CBD
PK Properties of CBD-NE compared to Epidyolex under Fasted Conditions | 0-24 hours
  Ratio of AUC0-24 to AUCinf for CBD, 7-OH-CBD and 7-COOH-CBD
Total Drug Exposure of CBD-NE compared to Epidyolex under Fed Conditions | 0-24 hours
  Sum of AUC0-24 of CBD, 7-OH-CBD and 7-COOH-CBD
Total Drug Exposure of CBD-NE compared to Epidyolex under Fasted Conditions | 0-24 hours
  Sum of AUC0-24 of CBD, 7-OH-CBD and 7-COOH-CBD
Total Drug Exposure of CBD-NE compared to Epidyolex under Fed Conditions | 0-24 hours
  Sum of AUCinf of CBD, 7-OH-CBD and 7-COOH-CBD
Total Drug Exposure of CBD-NE compared to Epidyolex under Fasted Conditions | 0-24 hours
  Sum of AUCinf of CBD, 7-OH-CBD and 7-COOH-CBD

OTHER OUTCOMES:
Comparison of PK Properties of CBD-NE under Fed and Fasted Conditions | 0-24 hours
  AUC0-24 for CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of PK Properties of Epidyolex under Fed and Fasted Conditions | 0-24 hours
  AUC0-24 for CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of PK Properties of CBD-NE under Fed and Fasted Conditions | 0-24 hours
  Cmax for CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of PK Properties of Epidyolex under Fed and Fasted Conditions | 0-24 hours
  Cmax for CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of PK Properties of CBD-NE under Fed and Fasted Conditions | 0-24 hours
  Tmax for CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of PK Properties of Epidyolex under Fed and Fasted Conditions | 0-24 hours
  Tmax for CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of PK Properties of CBD-NE under Fed and Fasted Conditions | 0-24 hours
  T1/2 for CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of PK Properties of Epidyolex under Fed and Fasted Conditions | 0-24 hours
  T1/2 for CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of PK Properties of CBD-NE under Fed and Fasted Conditions | 0-24 hours
  AUCinf of CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of PK Properties of Epidyolex under Fed and Fasted Conditions | 0-24 hours
  AUCinf for CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of PK Properties of CBD-NE under Fed and Fasted Conditions | 0-24 hours
  Ratio of AUC0-24 to AUCinf for CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of PK Properties of Epidyolex under Fed and Fasted Conditions | 0-24 hours
  Ratio of AUC0-24 to AUCinf for CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of Total Drug Exposure of CBD-NE under Fed and Fasted Conditions | 0-24 hours
  Sum of AUC0-24 of CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of Total Drug Exposure of Epidyolex under Fed and Fasted Conditions | 0-24 hours
  Sum of AUC0-24 of CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of Total Drug Exposure of CBD-NE under Fed and Fasted Conditions | 0-24 hours
  Sum of AUCinf of CBD, 7-OH-CBD and 7-COOH-CBD
Comparison of Total Drug Exposure of Epidyolex under Fed and Fasted Conditions | 0-24 hours
  Sum of AUCinf of CBD, 7-OH-CBD and 7-COOH-CBD
Assessment of 12-lead electrocardiogram (ECG) | 12 hours
  Change from pre-dose to 12 h in QRS interval as assessed by 12-lead ECG
Assessment of 12-lead electrocardiogram (ECG) | 12 hours
  Change from pre-dose to 12 h in heart rate as assessed by 12-lead ECG
Assessment of 12-lead electrocardiogram (ECG) | 12 hours
  Change from pre-dose to 12 h in PR interval as assessed by 12-lead ECG
Assessment of 12-lead electrocardiogram (ECG) | 12 hours
  Change from pre-dose to 12 h in QT interval as assessed by 12-lead ECG
Heart rate | 0-24 hours
  Change from pre-dose to post-dose in heart rate (beats per minute)
Blood pressure | 0-24 hours
  Change from pre-dose to post-dose in systolic and diastolic blood pressure (mm Hg)
Respiratory rate | 0-24 hours
  Change from pre-dose to 24 h in respiratory rate (breaths per minute)
Body Temperature | 0-24 hours
  Change from pre-dose to 24 h in body temperature (°C)
Composite Measure of Physical Abnormalities Observed in A Comprehensive Physical Exam | 12 hours
  Presence or absence of physical abnormalities in general appearance
Composite Measure of Physical Abnormalities Observed in a Comprehensive Physical Exam | 12 hours
  Presence or absence of physical abnormalities of ears
Composite Measure of Physical Abnormalities Observed in a Comprehensive Physical Exam | 12 hours
  Presence or absence of physical abnormalities of eyes
Composite Measure of Physical Abnormalities Observed in a Comprehensive Physical Exam | 12 hours
  Presence or absence of physical abnormalities of nose
Composite Measure of Physical Abnormalities Observed in a Comprehensive Physical Exam | 12 hours
  Presence or absence of physical abnormalities of throat
Composite Measure of Physical Abnormalities Observed in a Comprehensive Physical Exam | 12 hours
  Presence or absence of physical abnormalities of skin
Composite Measure of Physical Abnormalities Observed in a Comprehensive Physical Exam | 12 hours
  Presence or absence of physical abnormalities of chest
Composite Measure of Physical Abnormalities Observed in a Comprehensive Physical Exam | 12 hours
  Presence or absence of physical abnormalities of lungs
Composite Measure of Physical Abnormalities Observed in a Comprehensive Physical Exam | 12 hours
  Presence or absence of physical abnormalities of abdomen
Composite Measure of Physical Abnormalities Observed in a Comprehensive Physical Exam | 12 hours
  Presence or absence of physical abnormalities of lymph nodes
Composite Measure of Physical Abnormalities Observed in a Comprehensive Physical Exam | 12 hours
  Presence or absence of neurological abnormalities
Incidence of Adverse Events | minimum of 14 days, maximum of 28 days
  Number of participants with adverse events
Whole Blood Hemoglobin | 12 hours
  Change from pre-dose in whole blood hemoglobin (g/dL)
Whole Blood Hematocrit | 12 hours
  Change from pre-dose in whole blood hematocrit (%)
Whole Blood White Blood Cells | 12 hours
  Change from pre-dose in whole blood white blood cells (x10^3/uL)
Whole Blood Neutrophils | 12 hours
  Change from pre-dose in whole blood neutrophils (cells/uL)
Whole Blood Eosinophils | 12 hours
  Change from pre-dose in whole blood eosinophils (cells/uL)
Whole Blood Basophils | 12 hours
  Change from pre-dose in whole blood basophils (cells/uL)
Whole Blood Lymphocytes | 12 hours
  Change from pre-dose in whole blood lymphocytes (cells/uL)
Whole Blood Monocytes | 12 hours
  Change from pre-dose in whole blood monocytes (cells/uL)
Whole Blood Mean Platelet Volume | 12 hours
  Change from pre-dose in whole blood mean platelet volume (fL)
Whole Blood Platelet Count | 12 hours
  Change from pre-dose in whole blood platelet count (x10^9/L)
Whole Blood Red Blood Cell Count | 12 hours
  Change from pre-dose in whole blood red blood cell count (x10^6/uL)
Whole Blood Red Blood Cell Distribution Width | 12 hours
  Change from pre-dose in whole blood red blood cell distribution width (%)
Whole Blood Mean Corpuscular Volume | 12 hours
  Change from pre-dose in whole blood mean corpuscular volume (fL)
Whole Blood Mean Corpuscular Hemoglobin | 12 hours
  Change from pre-dose in whole blood mean corpuscular hemoglobin (pg)
Whole Blood Mean Corpuscular Hemoglobin Concentration | 12 hours
  Change from pre-dose in whole blood mean corpuscular hemoglobin concentration (g/dL)
Serum Sodium | 12 hours
  Change from pre-dose in serum sodium (mmol/L)
Serum Potassium | 12 hours
  Change from pre-dose in serum potassium (mmol/L)
Serum Chloride | 12 hours
  Change from pre-dose in serum chloride (mmol/L)
Serum Urea | 12 hours
  Change from pre-dose in serum urea (mg/dL)
Serum Creatinine | 12 hours
  Change from pre-dose in serum creatinine (umol/L)
Serum Estimated Glomerular Filtration | 12 hours
  Change from pre-dose in serum estimated glomerular filtration rate (mL/min/1.73^2)
Serum Total Protein | 12 hours
  Change from pre-dose in serum total protein (g/dL)
Serum Albumin | 12 hours
  Change from pre-dose in serum albumin (g/dL)
Serum Globulin | 12 hours
  Change from pre-dose in serum globulin (g/dL)
Serum Total Bilirubin | 12 hours
  Change from pre-dose in serum total bilirubin (mg/dL)
Serum Glucose | 12 hours
  Change from pre-dose in serum glucose concentration (mg/dL)
Serum Alanine Transaminase | 12 hours
  Change from pre-dose in serum alanine transaminase concentration (U/L)
Serum Aspartate Transaminase | 12 hours
  Change from pre-dose in serum aspartate transaminase concentration (U/L)
Serum Alkaline Phosphatase | 12 hours
  Change from pre-dose in serum alkaline phosphatase concentration (U/L)
Gamma Glutamyl Transferase | 12 hours
  Change from pre-dose in serum gamma glutamyl transferase concentration (U/L)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bier, MD, Principal Investigator — Apex Trials
Locations (1):
- Nutrasource Site (Apex Trials), Guelph, Ontario, Canada

REFERENCES:
- [Background] Legare CA, Raup-Konsavage WM, Vrana KE. Therapeutic Potential of Cannabis, Cannabidiol, and Cannabinoid-Based Pharmaceuticals. Pharmacology. 2022;107(3-4):131-149. doi: 10.1159/000521683. Epub 2022 Jan 28. PMID 35093949
- [Background] Devinsky O, Cross JH, Laux L, Marsh E, Miller I, Nabbout R, Scheffer IE, Thiele EA, Wright S; Cannabidiol in Dravet Syndrome Study Group. Trial of Cannabidiol for Drug-Resistant Seizures in the Dravet Syndrome. N Engl J Med. 2017 May 25;376(21):2011-2020. doi: 10.1056/NEJMoa1611618. PMID 28538134
- [Background] Knaub K, Sartorius T, Dharsono T, Wacker R, Wilhelm M, Schon C. A Novel Self-Emulsifying Drug Delivery System (SEDDS) Based on VESIsorb(R) Formulation Technology Improving the Oral Bioavailability of Cannabidiol in Healthy Subjects. Molecules. 2019 Aug 16;24(16):2967. doi: 10.3390/molecules24162967. PMID 31426272
- [Background] Huestis MA, Solimini R, Pichini S, Pacifici R, Carlier J, Busardo FP. Cannabidiol Adverse Effects and Toxicity. Curr Neuropharmacol. 2019;17(10):974-989. doi: 10.2174/1570159X17666190603171901. PMID 31161980
- [Background] Berl V, Hurd YL, Lipshutz BH, Roggen M, Mathur EJ, Evans M. A Randomized, Triple-Blind, Comparator-Controlled Parallel Study Investigating the Pharmacokinetics of Cannabidiol and Tetrahydrocannabinol in a Novel Delivery System, Solutech, in Association with Cannabis Use History. Cannabis Cannabinoid Res. 2022 Dec;7(6):777-789. doi: 10.1089/can.2021.0176. Epub 2022 Jul 5. PMID 35787693
- [Background] Taylor L, Gidal B, Blakey G, Tayo B, Morrison G. A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, Multiple Dose, and Food Effect Trial of the Safety, Tolerability and Pharmacokinetics of Highly Purified Cannabidiol in Healthy Subjects. CNS Drugs. 2018 Nov;32(11):1053-1067. doi: 10.1007/s40263-018-0578-5. PMID 30374683
- [Background] Abbotts KSS, Ewell TR, Butterklee HM, Bomar MC, Akagi N, Dooley GP, Bell C. Cannabidiol and Cannabidiol Metabolites: Pharmacokinetics, Interaction with Food, and Influence on Liver Function. Nutrients. 2022 May 21;14(10):2152. doi: 10.3390/nu14102152. PMID 35631293
- [Background] Britch SC, Babalonis S, Walsh SL. Cannabidiol: pharmacology and therapeutic targets. Psychopharmacology (Berl). 2021 Jan;238(1):9-28. doi: 10.1007/s00213-020-05712-8. Epub 2020 Nov 21. PMID 33221931
- [Background] Peng J, Fan M, An C, Ni F, Huang W, Luo J. A narrative review of molecular mechanism and therapeutic effect of cannabidiol (CBD). Basic Clin Pharmacol Toxicol. 2022 Apr;130(4):439-456. doi: 10.1111/bcpt.13710. Epub 2022 Feb 6. PMID 35083862
- See also: Approval for Epidiolex — https://www.newswire.ca/news-releases/jazz-pharmaceuticals-receives-health-canada-approval-for-epidiolex-r-cannabidiol-oral-solution-for-the-treatment-of-seizures-associated-with-three-rare-forms-of-epilepsy-830546952.html